CLINICAL TRIAL: NCT02124824
Title: Contribution of Endothelin-1 to Exercise Intolerance in HF
Brief Title: Contribution of Endothelin-1 to Exercise Intolerance in Heart Failure
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: F1418-P
Record Dates: First submitted 2014-02-11; First posted 2014-04-28 (Estimated); Results first posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — cyclo(Trp-Asp-Pro-Val-Leu)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Control (Experimental): Control
  Interventions: Drug: BQ-123
- Arm 2: Heart Failure (Experimental): Heart Failure
  Interventions: Drug: BQ-123

INTERVENTIONS:
Drug: BQ-123 — Endothelin subtype A antagonist

SUMMARY:
Heart disease is the leading cause of death in the United States, accounting for one in every four deaths in 2010 and costing over $300 billion annually in health care, medication, and lost productivity. Heart failure (HF), a clinical syndrome that develops as a consequence of heart disease, is characterized by the worsening of symptoms, such as dyspnea and fatigue, upon exertion, collectively defined as "exercise intolerance". Surprisingly, exercise intolerance does not correlate with the degree of cardiac contractile (ventricular) dysfunction, suggesting that changes in the peripheral circulation may be to blame for exercise intolerance in this cohort. Though there are a host of factors that may contribute to this impairment, disease-related increases in circulating endothelin-1 (ET-1) may be a significant factor in the sequelae of exercise intolerance in HF. Thus, the overall purpose of this Small Projects in Rehabilitation Research (SPiRE) proposal is to explore the contribution of ET-1 to chronic vasoconstriction in HF patients, and to examine whether inhibition of this pathway could improve vasodilatory ability, and thus exercise tolerance, in Veterans with HF.

DETAILED DESCRIPTION:
Specific Aim 1 will determine the direct effect of vascular endothelin-1 (ET-1) on skeletal muscle vasoconstriction in HF and age-matched controls. Intra-arterial infusion of the ETA subtype receptor will be undertaken to pharmacologically probe disease-related changes in the ET-1 pathway at rest and during exercise. It is hypothesized that ET-1-mediated vasoconstriction will be elevated in HF compared to controls at rest, such that ETA receptor blockade will augment blood flow in HF patients to a greater degree than age-matched controls. During exercise, the investigators anticipate that inhibition of the ETA receptor will augment skeletal muscle blood flow in HF patients compared to age-matched controls, leading to improved exercise tolerance and reduced skeletal muscle fatigue in this patient group. Specific Aim 2 will determine the potentiating effect of vascular endothelin-1 (ET-1) on sympathetic vasoconstriction in HF and age-matched controls. At rest, the investigators hypothesize that infusion of a sympathomimetic drug (norepinephrine, NE) will produce greater vasoconstriction in HF patients compared to age-matched controls, demonstrating a hypersensitivity of the alpha-adrenergic receptors. Inhibition of the ETA receptor will reduce "sensitivity" of NE-mediated vasoconstriction in HF patients towards that of age-matched controls, identifying ET-1 as a contributor to alpha adrenergic hypersensitivity in HF. During exercise, it is anticipated that NE-mediated vasoconstriction will be greater in HF patients compared to age-matched controls. Inhibition of the ETA receptor will reduce NE-mediated vasoconstriction during exercise. This will augment skeletal muscle blood flow, leading to improved exercise tolerance and reduced skeletal muscle fatigue in HF patients. The investigators anticipate that findings from the proposed work with ET-1 inhibition could thus provide a "missing link" of information in the investigators' understanding of skeletal muscle blood flow regulation and exercise tolerance in HF, ultimately leading to enhanced quality of life in this cohort.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion/Exclusion Criteria:

* The study group will include subjects with a history of stable cardiomyopathy (ischemic and non-ischemic, >3 months duration, ages 45-75 yrs) despite a minimum of 6 weeks of optimal treatment.
* Optimal therapy will be according to AHA/ACC and HFSA HF guidelines, including treatment with ACE and -blocker therapy (for at least 6 weeks), or have documented reason for variation, including medication intolerance, contraindication, patient preference, or personal physician's judgment.
* Patient enrollment will be limited to those individuals with NYHA class II and III symptoms, LVEF<35%, with no or minimal smoking history (<15 pk yrs), and without pacemakers.

Exclusion Criteria:

* Patients with atrial fibrillation or HF believed to be secondary to atrial fibrillation will be excluded.
* Patients with HF secondary to significant uncorrected primary valvular disease (except mitral regurgitation secondary to left ventricular dysfunction) will also be excluded.
* Patients will be sedentary, defined here as no regular physical activity for at least the prior 6 months and current activity level will be documented by an activity questionnaire.
* Patients must have no orthopedic limitations that would prohibit them from performing knee-extensor exercise.
* Due to the typical age of patients with HF, all women will be postmenopausal (either natural or surgical) defined as a cessation of menses for at least 2 years, and in women without a uterus, follicle stimulating hormone (FSH) >40 IU/L.
* Women currently taking hormone replacement therapy (HRT) will be excluded from the proposed studies due to the direct vascular effects of HRT Comorbidity Exclusion Criteria: Patients with significant non-cardiac comorbidities, which if present could alter the study results, will be excluded.

  * These include a diagnosis of Dementia
  * Severe COPD
  * Peripheral Vascular Disease
  * Anemia
  * Sleep-related Breathing Disorder
  * Severe Valvular Heart Disease
  * Diabetes (if on insulin therapy)
  * or End-stage Malignancy
* The investigators will also exclude morbidly obese patients (BMI >35), patients with uncontrolled Hypertension (>160/100), Anemia (Hgb<9) and Severe Renal Insufficiency (individuals with creatinine clearance <30 by the Cockcroft-Gault formula).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Wray, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Control | Arm 2: Heart Failure
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Control | Arm 2: Heart Failure | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (4) | 59 (6) | 62 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 1 | 1 | 2
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Blood Flow
Description: Ultrasound Doppler
Time Frame: two years
Measure: Mean (Standard Error); unit: ml/min
Arm/Group | Arm 1: Control | Arm 2: Heart Failure
Number analyzed (Participants) | 15 | 15
ml/min | 300 (50) | 275 (45)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Arm 1: Control | Arm 2: Heart Failure
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT02124824/Prot_SAP_000.pdf